CLINICAL TRIAL: NCT04085289
Title: A Randomized, Placebo-Controlled, Single-Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Galcanezumab in Healthy Chinese Subjects
Brief Title: A Study of Galcanezumab (LY2951742) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17057; I5Q-MC-CGAY (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Healthy
MeSH Terms: interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Galcanezumab (Experimental): Participants received single subcutaneous (SC) doses of 120 milligram (mg) or 240 mg Galcanezumab.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Participants received a single SC dose of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess how fast galcanezumab gets into the blood stream and how long it takes the body to remove it. Information about side effects will be collected. The study is open to healthy Chinese participants. It will last up to about 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are native Chinese (all 4 biological grandparents and both biological parents to be of Chinese origin)
* Participants who are overtly healthy males or females, as determined by medical history and physical examination

Exclusion Criteria:

* Participants who are currently enrolled in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Participants who have participated, within the last 30 days, in a clinical study involving an investigational product. If the previous investigational product has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed
* Participants who have received treatment with any CGRP (calcitonin gene related peptide) antibody (including galcanezumab), or antibody against CGRP receptor (including erenumab), or have received biologic agents (such as monoclonal antibodies) within 4 months or 5 half-lives (whichever is longer) prior to dosing
* Participants who have a history of multiple or severe allergies or has had an anaphylactic reaction to prescription or non-prescription drugs or food
* women who are lactating
* Participants who show evidence of positive human immunodeficiency virus antibodies, or positive hepatitis C antibody, or positive hepatitis B surface antigen, or active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- HuaShan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a single Subcutaneous (SC) dose of Placebo.
- 120 mg Galcanezumab SC: Participants received a single SC dose of 120 milligram (mg) Galcanezumab.
- 240 mg Galcanezumab SC: Participants received a single SC dose of 240 mg Galcanezumab.
Period: Overall Study
Arm/Group | Placebo | 120 mg Galcanezumab SC | 240 mg Galcanezumab SC
Started | 6 | 12 | 12
Received at Least One Dose of Study Drug | 6 | 12 | 12
Completed | 6 | 12 | 11
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 120 mg Galcanezumab SC | 240 mg Galcanezumab SC | Total
Number analyzed (Participants) | 6 | 12 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.70 (4.18) | 26.80 (6.03) | 28.80 (4.09) | 27.60 (4.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 4 | 8 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 12 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 12 | 12 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 6 | 12 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Galcanezumab
Description: Pharmacokinetics: Maximum Concentration (Cmax) of Galcanezumab.
Time Frame: 8, 24, 48, 96, 120, 168, 216, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2688, 3360 hours post-dose
Population: All randomized participants who received at least one dose of Galcanezumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | 120 mg Galcanezumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 12 | 12
micrograms per milliliter (μg/mL) | 12.6 (23) | 27.2 (23)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Galcanezumab
Description: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Galcanezumab.
Time Frame: 8, 24, 48, 96, 120, 168, 216, 264, 336, 504, 672, 1008, 1344, 1680, 2016, 2688, 3360 hours post-dose
Population: All randomized participants who received at least one dose of Galcanezumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day per milliliter(μg*day/mL)
Arm/Group | 120 mg Galcanezumab SC | 240 mg Galcanezumab SC
Number analyzed (Participants) | 12 | 12
micrograms*day per milliliter(μg*day/mL) | 558 (36) | 1190 (27)

ADVERSE EVENTS:
Time Frame: Baseline through Study Completion (Up To 20 weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 120 mg Galcanezumab SC | 240 mg Galcanezumab SC
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/12 | 1/12
Other Adverse Events (participants affected / at risk) | 5/6 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 120 mg Galcanezumab SC (N=12) | 240 mg Galcanezumab SC (N=12)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=6) | 120 mg Galcanezumab SC (N=12) | 240 mg Galcanezumab SC (N=12)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 1 (2)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (6) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Bacterial test (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 3 (8)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil percentage increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 2 (2)
Urinary casts present (Investigations) | 1 (1) | 0 (0) | 2 (3)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/2 (0) | 1/4 (1) | 0/1 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04085289/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT04085289/SAP_001.pdf